CLINICAL TRIAL: NCT02025452
Title: Rapid Diagnostics and Probiotic Therapy for Paediatric Acute Gastroenteritis - a Randomized, Factorial, Controlled, Placebo-controlled, Pilot Trial
Brief Title: Novel Diagnostics and Probiotics to Improve Management of Paediatric Acute Gastroenteritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jeffrey Pernica (Other)
Collaborators: Grand Challenges Canada (Other); BioGaia AB (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey Pernica, Head, Division of Pediatric Infectious Disease, Hamilton Health Sciences Corporation
Organization: Hamilton Health Sciences Corporation (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HHS 13-749
Record Dates: First submitted 2013-12-28; First posted 2014-01-01 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Acute Gastroenteritis
Keywords: diarrhoea; gastroenteritis; rapid diagnostics; probiotics; sub-Saharan Africa
MeSH Terms: conditions — Diarrhea; Gastroenteritis | interventions — Rapid Diagnostic Tests; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rapid diagnostics and probiotic (Active Comparator)
  Interventions: Other: Rapid diagnostic; Dietary Supplement: Probiotic
- Rapid diagnostics and placebo (Placebo Comparator)
  Interventions: Other: Rapid diagnostic; Other: Placebo
- Delayed diagnostics and probiotic (Experimental)
  Interventions: Dietary Supplement: Probiotic
- Delayed diagnostics and placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Rapid diagnostic — Specimens from rectal mucosa will be obtained using flocked swabs at enrolment. Those in 'rapid diagnostic' groups will have them tested using multiplex PCR the day of enrolment and participants with treatable pathogens will have antimicrobials provided. Those in 'delayed diagnostic' groups will have the swabs batched at tested at the conclusion of the study, being treated as per standard of care.
  Arms: Rapid diagnostics and placebo; Rapid diagnostics and probiotic
Dietary Supplement: Probiotic — Lactobacillus reuteri suspended in vegetable oil, 5 drops/day (1 x 10e8 CFU) x 2 months
  Arms: Delayed diagnostics and probiotic; Rapid diagnostics and probiotic
Other: Placebo — Identical in appearance to L. reuteri probiotic (same bottle), but simply vegetable oil. Dose is 5 drops/day x 2 months.
  Arms: Delayed diagnostics and placebo; Rapid diagnostics and placebo

SUMMARY:
Many children admitted to hospital in Botswana without bloody diarrhoea are presumed to have viral gastroenteritis and so not treated with antibiotics - but they may indeed have a treatable cause for their illness. We will conduct a randomized trial to see if rapid testing using novel methods to identify potentially treatable causes of diarrhoea leads to improved outcomes. We will also be randomizing children to probiotic therapy versus placebo (the standard of care) to see if this treatment decreases the duration of diarrhoea. The proposed study is a pilot trial, necessary before embarking on a large multi-centre trial.

ELIGIBILITY:
Inclusion Criteria:

* acute non-bloody gastroenteritis

Exclusion Criteria:

* diarrhoea > 14 days
* sepsis, pneumonia, UTI, meningitis requiring empiric antibiotic therapy
* malignancy, IBD
* known link to another patient with diarrhoea of defined aetiology
* transferred in already on antimicrobials
* live outside study area
* children with severe acute malnutrition will be eligible for diagnostic arm but not probiotic arm

Ages: 2 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Height z-score (HAZ) adjusted for initial HAZ | 60 days post-enrollment

SECONDARY OUTCOMES:
mortality | 60 days post-enrollment
environmental enteropathy score | 60 days post-enrollment
duration of diarrhoea | estimated average duration ~ 4 days.
  Note that presence of diarrhoea will be checked daily during admission. Total duration of diarrhoea will be verified with the caregiver by telephone 7 days after the participant was discharged home.
Weight z-score (WAZ) adjusted for initial WAZ | 60 days after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Pernica, MD, Principal Investigator — McMaster University
Locations (3):
- Botswana (3):
  - Princess Marina Hospital, Gaborone
  - Scottish Livingstone Hospital, Molepolole
  - Bamalete Lutheran Hospital, Ramotswa